CLINICAL TRIAL: NCT05341453
Title: The Effect of Intensive Hippotherapy on the Psychomotoric Development of Children With Spinal Muscular Atrophy
Brief Title: Hippotherapy in Children With Spinal Muscular Atrophy
Acronym: HIPOSMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kamila Řasová, assoc. prof. PhDr. Kamila Řasová, Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18032022
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Spinal Muscular Atrophy
Keywords: hippotherapy; children; psychomotor development; physiotherapy; quality of life; posture; motor skills; therapeutic riding; muscle fatigue
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial. 16 children will be randomized into two interventional groups, on classic physiotherapy, the second hippotherapy. Participants both groups will undergo 12 therapies, twice a day, 15 minutes long. Before and in 6 day all children will be examined by a blinded independent clinician.
Who Masked: Outcomes Assessor
Masking Description: All participants of the study will undergo a clinical examination including a questionnaire survey, led by a blinded independent examiner, who will not have access to intervention documentation. The examiner will see each patient twice, before the first intervention and 6 days later in the end last therapy. The examiner will be prohibited to talk about the therapy attended. The parents of patients will be informed about the character of the examination ant the importance of the most objectivity possible. All therapists can apply both interventions, therefore masking is more efficient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individual physiotherapy (SMA-SOC) (Active Comparator): Individual physiotherapy will be performed according to the recommended SMA-SOC guidelines.
  Interventions: Procedure: Individual physiotherapy (SMA-SOC)
- Hippotherapy by the children with cerebral palsy (Experimental): Hippotherapy by the children with cerebral palsy is an accredited form of hippotherapy, whose methodology is based on the clinical picture of cerebral palsy, but its procedures are applicable to a wider group of children with disabilities. Therefore, investigators assume its effect for children with SMA.
  Interventions: Procedure: Hippotherapy
- Therapeutic grooming (Other): In order to influence the psychomotor development in a comprehensive way, the psychosocial activity of therapeutic grooming will also be included in the study. Its goal is to support children's communication, their interaction with the environment, the ability to establish contact with the horse and the overall emotional support of children with SMA.
  Interventions: Procedure: Therapeutic grooming

INTERVENTIONS:
Procedure: Individual physiotherapy (SMA-SOC) — Therapeutic procedures according to the recommended standard (SMA-SOC) will be used in the therapy. Elements of breathing gymnastics, vibration techniques, stretching, eccentric and concentric exercise procedures will be combined. Individual physiotherapy will be conducted on the basis of set goals from the kinesiological examination, it will be adapted to the individuality of the child - his cooperation, fatigue and sleep time.
  Arms: Individual physiotherapy (SMA-SOC)
Procedure: Hippotherapy — HT by CP is an accredited form of hippotherapy, whose methodology is based on the clinical picture of cerebral palsy, but its procedures are applicable to a wider group of children with disabilities. Therefore, investigators anticipate it´s effect for children with SMA.
  Based on a special type of examination, this method precisely determines the "type / breed" of the horse according to the biomechanics of the movement of its back in the step, the position of the child and the neurophysiological function of the back - differentiation or sensorimotor skills. Furthermore, according to the course of therapy, the physiotherapist determines the pace of the horse's step, its length, selects special manual contacts according to the current situation and adjusts the duration of therapy to the client's fatigue.
  Therapy will be performed by therapists with professional competence to perform hippotherapy by children with CP.
  Other Names: Hippotherapy by the children with cerebral palsy (HT by CP)
  Arms: Hippotherapy by the children with cerebral palsy
Procedure: Therapeutic grooming — In order to influence the psychomotor development in a comprehensive way, the psychosocial activity of therapeutic grooming will also be included in the study. Its goal is to support children's communication, their interaction with the environment, the ability to establish contact with the horse and the overall emotional support of children with SMA. The purpose of this activity is to clean the horse, its possible guide, stroking and contact with the horse, work from the ground.
  Arms: Therapeutic grooming

SUMMARY:
The randomized controlled trial is aimed to discover the physiotherapy and hippotherapy effect and efficacy on children with SMA. The concept is to utilized two types of physiotherapy - the first concept is classic physiotherapy and the second one is hippotherapy. The hippotherapy concept will be in intervals of 15 minutes twice a day, the physiotherapy will be in intervals of 30 minutes once a day. In-patient therapy will be for 6 days. The efficacy will be assessed by biomedical measures - Qualisys Motion Capture Systems 2020.3., by molecular biological markers (lncRNA) in blood and by surface electromyography (EMG). The primary goal of this study is to compare two physiotherapeutic approaches - the recommended form of classical physiotherapy and the method on a neurophysiological basis - hippotherapy. The secondary intention of the research will be the appropriate intensity of therapy so that unwanted muscle fatigue does not occur.

DETAILED DESCRIPTION:
Spinal muscular atrophy is rare neuromuscular disease, it is caused by gene mutation survival motor neuron 1 (SMN1). This gene encodes survival motor neuron(SMN) protein. This protein is most important to survive alfa-motoric neurons in spinal cord. When this protein doesn´t work, no signals go from brain to skeletal muscles and fazic muscles of body. In the end weakening breathing muscles and internal organs muscles. The first treatment is pharmacological treatment. There is a lot of research about medicament treatment, the famous treatment in Czech Republic is medicine Spinraze and from year 2020 medicine Zongelsma. This, however, more often puts more difficulty on complex rehabilitation. An empirical observation has found out that complex rehabilitation has positive effect on progress of disease and on self-sufficiency of people and children with SMA. Physiotherapy is one of the recommended rehabilitation types.

The use of rehabilitation procedures is common in clinical practice. In a 2016 study, 105 adults with SMA were asked how many of them used physiotherapy. A total of 86% of respondents received these services, yet the authors of the article conclude that further research is needed to understand the impact of physiotherapy in SMA.

Nevertheless, there is a lot of discussion if physiotherapy is really good for people and children with SMA. Some research shows us, that physiotherapy doesn´t worsen this disease. Researchers showed that strength training 3 times a week does not show side effects in children under 10 years of age, in some cases trends in improving muscle strength and motor functions have been observed.

Because in physiotherapy therapists work primarily with muscles, and a lot of activity can cause fatigue of skeletal muscles and worsen their function. But from clinical work scientists know that the effect of physiotherapy is extensive. There is a research on mice which shows the effect of physiotherapy on the strength activities and the aerobic activities.

Research to better elucidate the intensity of physiotherapy has not yet been published. Motes et al. monitored a total of 16 patients with SMA aged 10 - 55 years, who regularly underwent home autotherapy for 16 months - cycling and strengthening. The authors did not find any side effects of exercise on strength, function or fatigue during the study. However, the oxidation capacity has been reduced and according to the authors, further research is needed in this area.

In the United States, the "Standard of Care" (SMA-SOC) has been developed for SMA, which regulates the rehabilitation care of children and adults with SMA according to the degree of mobility. In the framework of the said directive, the stretching of contractures, swimming, water therapy, light strength exercises and a verticalization stand are recommended within the framework of physiotherapy, and horse riding is also mentioned - but without more detailed information. Vibration techniques and positioning are recommended to improve breathing. Recommended exercises for seated persons also include concentric and eccentric exercises and aerobic and general fitness exercises with and without resistance. According to the directive, the duration of therapy should be adapted to the individual patient. For walkers, the exercise program may include some forms of balance exercises, dynamic and static.

In a study from 2021, physiotherapists were asked about their knowledge of SMA-SOC and its use in practice. Most of them stated that after individuals with SMA started disease-modifying pharmacotherapy, they would recommend increasing the frequency and duration of therapeutic interventions. The authors agree that in practice there are differences in the care of people with SMA, especially in the frequency and duration of specific interventions. At the same time, they state that these findings can identify future research needs and thus extend SMA-SOC to rehabilitation management best practices.

Our goal is to compare two physiotherapeutic approaches - the recommended form of classical physiotherapy and the method on a neurophysiological basis - hippotherapy. Due to the nature of the disease, investigators expect a greater effect in the method of Hippotherapy in cerebral palsy (CP), where several muscle chains work simultaneously and thus succeeds in activating weakened muscles within the chain, which eliminates possible fatigue and worsening of the condition. However, investigators also expect a positive effect in the recommended form of classical physiotherapy. Here, however, due to the lower intensity of the sensory environment and the possible complexity of movement, investigators assume less effectiveness than hippotherapy.

The secondary intention of the research will be the appropriate intensity of therapy so that unwanted muscle fatigue does not occur. Investigators will therefore investigate the neurophysiological mechanisms of rehabilitation that investigators will monitor using long non-coding RNAs (lncRNAs) involved in important cellular regulation, including regulation of genomic imprinting, epigenetic chromatin modification, transcriptional interference, and nuclear export. The lncRNA, SMN-antisense 1 (SMN-AS1), has been shown to repress the expression of the duplicate survival motor neuron 2 (SMN2) gene by binding Polycomb repressive complex 2 (PRC2) to its locus. Increasing the transcriptional activity of an almost identical SMN2 gene can functionally compensate for the loss of SMN1, increase the amount of SMN protein and thus improve the prognosis of the disease. Chemically modified oligonucleotides have been proposed that disrupt the interaction between SMN-AS1 and PRC2, which inhibits the action of PRC2 and thus leads to increased SMN2 expression. Investigation of lncRNAs involved in the processes of gene regulation of these genes may help to understand the neurophysiological effects of rehabilitation of children with SMA.

ELIGIBILITY:
Inclusion Criteria:

* clinic diagnosis SMA (I, II, and III types)
* no changing medicine 6 months at least
* without another grave diseases

Exclusion Criteria:

* hip subluxation
* allergies to horses and the environment of horse stables
* insurmountable fear of the horse

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-10-22 (Estimated); Study Completion 2025-10-22 (Estimated)

PRIMARY OUTCOMES:
The ability of the thorax to change shape | 15 minutes
  The examination will take place lying on your back. 3 position markers will be placed on each side of the thorax, in the area of the distal end of the sternum axes, at the level of the 3rd rib and at the lowest arch of the 10th rib. Their position during exhalation and inspiration will be measured, and the change in thorax circumference will be evaluated. The aim of this test is to objectify the change in respiratory stereotype. After therapy, investigators expect a greater ability of the thorax to change direction.
Sitting symmetry | 5 minutes
  Observations will be made by sitting on a therapy cylinder. There will be special markers on the body (on clothes) of children: lower angles of the scapulae axes, ridge of the iliac axes, sacroiliac joint (SI) on both sides and in the area of the L4 vertebra and navel. Investigators will measure the symmetry of these marks in each other's position and the movement in which the child will walk back and forth with his hands. Markers will be analyzed using Qualisys Motion Capture Systems 2020.3. Acceleration and change of position will be evaluated in the second time.
Work with the center of gravity | 10 minutes
  Observation will be performed by sitting on therapeutic cylinder. 3 position markers will be used on each side of the body, at the root of the palm, in the area of the SI joint and at the level of the temporomandibular joint. The change of markers will be measured from the starting position until the child is stretched to the side (torso tilt with lug) and forward (torso flexion with forearm). The monitoring child will be motivated to reach for the toy. The goal is to evaluate the stability of children. Investigators assume, that after therapy investigators can see better work with the center of gravity.
Muscle fatigue | 10 minutes
  Investigators will measure muscle fatigue after physical activity using surface EMG. The child will lie on his back, therapist will provide a toy in the area of his opposite knee. The child will stretch for a toy. This act will be 30 s. Investigators will evaluate activity m.obliquus externus abdominis at the beginning and end of this specific activity. Goal is to evaluate muscle fatigue. Investigators assume, that after intensive therapeutic program will be muscle fatigue lower.
Hammersmith function scale for children with spinal muscular atrophy | 40 minutes
  The examination will follow a standardized procedure. The maximum score of the standardized test is 64 points on each side, the minimum is 0 points. A higher score means an improvement in the child's movement possibilities.
Deep neck flexor endurance test | 5 minutes
  The examination will follow a standardized procedure. Longer holding in the position means a better result, the exact holding time is not standardized for this test.
Neck extensor endurance test | 5 minutes
  The examination will follow a standardized procedure. Longer holding in the position means a better result, the exact holding time is not standardized for this test.
Spirometric measure | 2 minutes
  The spirometer will be used to determine the forced expiratory volume in 1 second forced expiratory volume at one second (FEV1) value, i.e the volume of air exhaled after the maximum inspiration with the greatest effort within 1 second. The change in value at the beginning and end of the rehabilitation stay will be evaluated.

SECONDARY OUTCOMES:
Quality of life assessment | 120 minutes
  Parents of child with SMA will fill special questionnaire at the beginning and 4-5 weeks after end of the rehabilitation. The ICF score set, more precisely the ICF-based Documentation Form, the category Children with cerebral palsy Brief (below 6 years old),supplemented by some items from the basic rehabilitation set, will be used to evaluate the quality of life.
Monitoring of molecular biological indicators of rehabilitation | 10 minutes
  Samples treated in this way can be safely stored at room temperature for longer periods of time (up to three days or more). Blood samples stored in Ribonucleic acid (RNAlater)® Solution achieve RNA quality comparable to the quality of samples processed immediately according to commercial websites. The expected average total RNA yields will be about 2-4 /g / 0.5 ml all blood. Total RNA will be transcribed into complementary deoxyribonucleic acid complementary (cDNA) by reverse transcriptase. To avoid error, the expression of human lncRNA and internal endogenous gene (e.g., GAPDH) will be quantified using RNA obtained from blinded samples (i.e., concealment of sample origin allocation).

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Rasova, as.prof.Dr., Study Director — Clinic of rheumatology and rehabilitation, Third medical faculty CU and Faculty Thomayer Hospital
Locations (1):
- Kamila Řasová, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Clinical Study Report (CSR) and Analytic Code will be shared when data is collected.
  Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF) are shared as attachment of this registration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Done now: Study protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF) 22.4. - 29.4.2022, 24.9. - 30.9.2022: Clinical Study Report (CSR) 2023 - 2024: Analytic Code
Access Criteria: Researcher can write us for access to data code.
URL: https://www.chmirakl.cz/

REFERENCES:
- Available data/document: Study Protocol — https://www.chmirakl.cz/aktuality/study-protokol
- Available data/document: Statistical Analysis Plan — https://www.chmirakl.cz/aktuality/statistical-analysis-plan
- Available data/document: Informed Consent Form — https://www.chmirakl.cz/aktuality/type-informed-consent-form

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT05341453/Prot_SAP_000.pdf